CLINICAL TRIAL: NCT03722043
Title: Investigating the Impact of A Veteran-Focused Parenting Program on Parenting Stress, Competence and Parenting Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Lisa Cromer, Associate Professor, University of Tulsa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TU1726
Record Dates: First submitted 2017-08-18; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Parenting; Military Family

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenting Program (Experimental): All study participants will receive our parenting program curriculum. There will not be a control group.
  The parenting program will include the topics of mindful parenting strategies, emotional regulation, positive discipline, and positive parenting/attachment. Participants will be provided skills to develop strategies for each of the modules. Each session will contain elements of group troubleshooting and practice in-session. Practice at home will be assigned so that participants can continue to practice and implement these skills and strategies in their homes.
  The program is taken from a published, empirically based program called "Everyday Parenting: A Professional's Guide to Building Family Management Skills" written by Thomas Dishion, Elizabeth Stormshak, and Kathryn Kavanagh.
  Interventions: Behavioral: Parenting Program

INTERVENTIONS:
Behavioral: Parenting Program — Parents will participate in a 5-week parenting program designed to uniquely work with veteran families. The program will target the following areas: mindful parenting strategies, emotional regulation, positive discipline, positive parenting/attachment, and sleep.

SUMMARY:
Veterans or spouses of veterans with a minor child will participate in a five-week parenting program. The goals of the parenting program are to assist in improving parent's sense of competence, improving parent's emotional regulation abilities, and lower parental stress by incorporating mindfulness and values-based parenting principles. The program will utilize evidence-based practices that will be delivered in a manner that incorporates aspects of military culture (i.e., language and concepts are tailored to that used within military culture). Mindfulness and acceptance and commitment therapy have been shown to be effective in treating service members [1], and this will be the first study that examines how learning these principles do or do not impact parenting stress, competence, and practices. The parenting program is free, and is offered by the investigators as a community service. Participation in the parenting program does not obligate enrollment in the research study.

DETAILED DESCRIPTION:
There are over 312,000 Veterans living in the state of Oklahoma [2]. The Coffee Bunker is a non-profit community agency in Tulsa, Oklahoma that serves as the flagships program for Serving Our Service Members (S.O.S). The Coffee Bunker's mission is to offer support to service members and Veterans by helping them reintegrate back into their families and communities. The overall purpose of the present study is to work with the Coffee Bunker in offering support towards their mission, specifically in delivering organized parenting programs to service members and Veterans.

Challenges of reintegration after a military deployment can increase levels of stress for Veterans, spouses, and their children. In fact, it is common for Veterans or service members who struggle with reintegration in their family to report feelings of isolation and lack of perceived control, which may impact their ability to parent effectively. The struggles of parents can negatively impact the functioning of the family, such that children may exhibit more behavioral problems and Veterans parents may be more vulnerable to mental health symptomology [3, 4]. Fortunately, research suggests that positive and effective parenting practices can mitigate family stressors [5, 6]. As such, given the stressors of reintegration among military families, it may be advantageous to implement an evidence-based psychoeducation parenting program tailored to Veterans. The goals of the parenting program are to assist in improving parent's sense of competence, improving parent's emotional regulation abilities, and lower parental stress. The current project will be evaluating possible benefits from an evidence-based parenting program with military families. The parenting program is free, and is offered by the investigators as a community service. Participation in the parenting program does not obligate enrollment in the study. This is made possible by one of the PI's (Zanotti's) Schweitzer Fellowship; Zanotti is conducting the parenting program along with Dr. Cromer, as a community service.

The research portion of this study will be voluntary, and while participants will be recruited from the parenting program, it will be made clear that they can opt into the parenting program without doing any of the research measures. The research portion evaluates whether participation in the parenting program reduces parenting stress, increases feelings of parenting competence, and improves parenting practices. This study is unique in that evidence-based practices will be delivered in a manner that incorporates aspects of military culture (i.e., language and concepts are tailored to that used within military culture). The parenting program will incorporate mindfulness and values-based parenting principles. Mindfulness and acceptance and commitment therapy have been shown to be effective in treating service members [1] and this will be the first study that examines how learning these principles do or do not impact parenting stress, competence, and practices.

ELIGIBILITY:
Inclusion Criteria:

* Must be a parent of a minor
* Must be fluent in English
* Must be a veteran or have a spouse who is a veteran

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-08 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Parenting Sense of Competence after 6 weeks, using the Parenting Sense of Competence Scale (PSOC; Johnston & Marsh, 1989) | Pre-treatment, post-treatment (i.e., approximately 6 weeks after the start of the parenting program).
  The PSOC consists of 16 items about parents' confidence on being a parent, answered on a six-point scale ranging from ''strongly disagree'' to ''strongly agree''. Scoring for some items is reversed so that, for all items, higher scores indicate greater parenting self-esteem. Two subscales measure efficacy (seven items) and satisfaction (nine items) in parenting.

SECONDARY OUTCOMES:
Change in Parenting Stress after 6 weeks, using the Parenting Stress Scale (PSS; Berry & Jones, 1995) | Pre-treatment, post-treatment (i.e., approximately 6 weeks after the start of the parenting program)
  This 18-item self-report measure assesses common stressors and positive components associated with parenting. Items are rated on a five-point Likert scale (i.e., 1=strongly disagree, 5=strongly agree). Positive items are reverse scored. A total stress score is generated by summing the items together (i.e., range=18-90). Higher scores indicate greater parental stress.
Change in Parent's Emotion Regulation Abilities after 6 weeks, using the Difficulties in Emotion Regulation Scales (DERS; Gratz & Roemer, 2004) | Pre-treatment, post-treatment (i.e., approximately 6 weeks after the start of the parenting program)
  This 36-item questionnaire assesses aspects of emotion regulation and dysregulation strategies utilized by individuals. Items are rated on a five-point Likert scale (i.e., 1=almost never, 5=almost always). Negatively worded items are reverse scored. Six component scores as well as a total scare is generated. Higher scores indicate greater emotion dysregulation.
Change in Parenting Practices after 6 weeks, using the Parenting Practices Interview (PPI; Webster-Stratton, Reid, & Hammond, 2001) | Pre-treatment, post-treatment (i.e., approximately 6 weeks after the start of the parenting program)
  The PPI was adapted from the Oregon Social Learning Centre's Discipline Questionnaire. Two subscales were used; Harsh Discipline (14 items, a 1⁄4 0.79), and Positive Parenting (15 items, a 1⁄4 0.67). Parents reported the probability and the frequency with which they used the different strategies on a seven-point scale.
Change in Parenting Styles after 6 weeks, using the Alabama Parenting Questionnaire-Short Form (APQ-9; Elgar, Waschbusch, Dadds, & Sigvaldason, 2007) | Pre-treatment, post-treatment (i.e., approximately 6 weeks after the start of the parenting program)
  This 9-item self-report measure assesses three styles of parenting: positive parenting, inconsistent discipline, and poor supervision. It has good convergent validity with longer measures of parenting styles. Responses are provided on a Likert scale where 1 = never, 2 = almost never, 3 = sometimes, 4= often, and 5 = always.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cromer, PhD, Study Chair — University of Tulsa
Locations (1):
- Coffee Bunker, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Vujanovic, A. A., Niles, B., Pietrefesa, A., Schmertz, S. K., & Potter, C. M. (2013). Mindfulness in the treatment of posttraumatic stress disorder among military veterans. Professional Psychology: Research and Practice, 42, 24-31.
- [Background] United States Census Bureau. (2015). Veteran Statistics-Oklahoma. Retrieved from https://www2.census.gov/library/infographics/2015/comm/vets/ok-vets.pdf.
- [Background] Lester P, Peterson K, Reeves J, Knauss L, Glover D, Mogil C, Duan N, Saltzman W, Pynoos R, Wilt K, Beardslee W. The long war and parental combat deployment: effects on military children and at-home spouses. J Am Acad Child Adolesc Psychiatry. 2010 Apr;49(4):310-20. PMID 20410724
- [Background] Louie, A. D., & Cromer, L. D. (2014). Parent-child attachment during the deployment cycle: Impact on reintegration parenting stress. Professional Psychology: Research and Practice, 45(6), 496.
- [Background] Lester, P., & Bursch, B. (2011). The long war comes home: Mitigating risk and promoting resilience in military children and families. Psychiatric Time, 28(7), 26-29.
- [Background] Veltman, M. W., & Browne, K. D. (2001). Three decades of child maltreatment research implications for the school years. Trauma, Violence, & Abuse, 2(3), 215-239.
- [Result] Johnston, C., & Mash, E. J. (1989). A measure of parenting satisfaction and efficacy. Journal of Clinical Child Psychology, 18(2), 167-175.
- [Result] Berry, J. O., & Jones, W. H. (1995). The parental stress scale: Initial psychometric evidence. Journal of Social and Personal Relationships, 12, 463-472.
- [Result] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Result] Webster-Stratton C, Reid MJ, Hammond M. Preventing conduct problems, promoting social competence: a parent and teacher training partnership in head start. J Clin Child Psychol. 2001 Sep;30(3):283-302. doi: 10.1207/S15374424JCCP3003_2. PMID 11501247
- [Result] Elgar, F. J., Waschbusch, D. A., Dadds, M. R., & Sigvaldason, N. (2007). Development and validation of a short form of the Alabama Parenting Questionnaire. Journal of Child and Family Studies, 16(2), 243-259.